CLINICAL TRIAL: NCT03264573
Title: Role of Stem Cells, Platelet Rich Plasma and Combination of Them in Treatment of Scars
Brief Title: Role of Stem Cells, Platelet Rich Plasma in Treatment of Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heba Mohamed Saad Eldien (Other)
Collaborators: M.A. Eloteify (Unknown); Ahmed Kamal Osman (Unknown); G.M. Hafsa (Unknown)
Responsible Party: Sponsor-Investigator, Heba Mohamed Saad Eldien, Professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSCs, PRP, Scar
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Atrophic Scar
Keywords: Atrophic scar; PRP; ADSCs

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stem cell, PRP (Active Comparator): Adipose derived MSCs, versus Platelet rich plasma
  Interventions: Biological: Stem cell; Device: MSCs
- Stem cell, Stem cell and PRP (Active Comparator): Adipose derived MSCs alone, other group is injected Adipose derived MSCs, and Platelet rich plasma
  Interventions: Biological: Stem cell; Device: MSCs

INTERVENTIONS:
Biological: Stem cell — after scar revision PRP is injected intradermally, also adipose derived mesenchymal stem cells
  Other Names: PRP
Device: MSCs — manual separation of platelets rich plasma and undifferentiated mesenchymal stem cells
  Other Names: Stem cell and PRP

SUMMARY:
The Objectives of this randomized controlled trial aiming to establishing a protocol of post scar revision care and to Study the effect of PRP and/or Adipose derived Mesenchymal Stem cell injection in improvement of atrophic scar after scar revision.

DETAILED DESCRIPTION:
Forty patients with atrophic scar since one to five years including 25 males and 15 females with ages ranging from ten to 35 years with main age of 22.68 will be divided into four groups each included ten patients. One group will be treated with scar revision only (control group or group I), 2nd group will be injected with PRP after scar revision, 3rd group will be injected with ADSCs after scar revision and the 4th group will be injected with a combination of PRP and ADSCs after scar revision. All groups were assisted pre-operative and six months post-operative. Complications, Scar width, Vancouver scar scale (VSS), surgeon assessment scar scale and patient assessment scar scale will be considered the outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patient with atrophic scar.
* Age group: 5 years up to 35 years.
* No previous medications, surgeries or laser therapy.

Exclusion Criteria:

* Patient with hypertrophic or pigmented scar.
* Patient with any blood disease.
* Patients with lipodystrophy.

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction (Patient Assessment Scar Scale) | 6 months
  Patient Assessment Scar Scale

SECONDARY OUTCOMES:
Doctor satisfaction (Vancouver Scar Scale) | 6 months
  Vancouver Scar Scale (VSS)